CLINICAL TRIAL: NCT00763529
Title: Elocon vs Fluticasone in Localized Psoriasis
Brief Title: Elocon vs Fluticasone in Localized Psoriasis (P03197)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03197
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Mometasone Furoate; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Mometasone
- Arm 2 (Active Comparator)
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Mometasone — Mometasone furoate cream 0.1% applied once daily
  Other Names: Elocon; SCH 32088
  Arms: Arm 1
Drug: Fluticasone — Fluticasone propionate cream 0.05% applied twice daily
  Other Names: Cutivate
  Arms: Arm 2

SUMMARY:
This is an open-label, randomized, parallel-group clinical study. The primary objective is to assess the difference in response rate between mometasone furoate cream 0.1% (once daily) vs fluticasone propionate cream 0.05% (twice daily) by the end of Day 4 and Day 8 in the management of Indian patients with localized psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* Written informed consent
* Having localized psoriasis (not more than 5-6 patches)
* Total size of all patches should be below 8" x 8"
* Each patient should exhibit any of the following 4 signs of dermatoses:

  * erythema
  * palpability
  * scaling
  * itching (pruritus)

Each of the above signs would be grades according to the following scale:

0 = none

1. = slight
2. = moderate
3. = severe The total Disease Severity Score (ie, the sum of the scores for each of the signs) should be at least 6 (indicative of a moderate to severe disease status)

Exclusion Criteria:

* Pregnancy or lactation
* Hypersensitivity to any of the components of the test medication
* Signs of atrophy in the target area
* Lesions on palms, soles, and scalp
* Individuals who may require medications that might affect the natural course of the disease
* Not having used systemic corticosteroids or antimetabolites or any other topical corticosteroid within 2 weeks prior to enrollment in the study
* Concomitant tuberculosis/viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2005-01-01 (Actual); Study Completion 2005-01-01 (Actual)

PRIMARY OUTCOMES:
Reduction in mean symptom scores for erythema, induration, pruritus, and scaling on Day 4. | Day 4
Reduction in mean symptom scores for erythema, induration, pruritus, and scaling on Day 8. | Day 8
Clinical evaluation of the change in disease status which would be defined as improvement by Day 4 relative to their severity at entry in treated areas. | Day 4
Clinical evaluation of the change in disease status which would be defined as improvement by Day 8 relative to their severity at entry in treated areas. | Day 8

SECONDARY OUTCOMES:
Reduction in mean symptom scores for erythema, induration, pruritus, and scaling on Day 15. | Day 15
Reduction in mean symptom scores for erythema, induration, pruritus, and scaling on Day 22. | Day 22
Reduction in mean symptom scores for erythema, induration, pruritus, and scaling on Day 29. | Day 29
Clinical evaluation of the change in treated areas relative to their severity at entry would also be evaluated on Day 15. | Day 15
Clinical evaluation of the change in treated areas relative to their severity at entry would also be evaluated on Day 22. | Day 22
Clinical evaluation of the change in treated areas relative to their severity at entry would also be evaluated on Day 29. | Day 29